CLINICAL TRIAL: NCT02852109
Title: Diffusion Tensor Imaging to Judge the Prognosis of Patients With Diffuse Axonal
Brief Title: Diffusion Tensor Imaging to Judge the Prognosis of Patients With Diffuse Axonal Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaoqiang Wang, Associate chief physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-009
Record Dates: First submitted 2016-04-15; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Diffuse Axonal Injury
MeSH Terms: conditions — Diffuse Axonal Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- experimental group: patients who was firstly diagnosed as diffuse axonal injury
- control group: patients negative for magnetic resonance examination with no trauma

SUMMARY:
The investigators will examine 15 patients who was firstly diagnosed as diffuse axonal injury and 15 patients negative for magnetic resonance examination with no trauma with DTI(diffusion tensor imaging). The investigators then determine the FA（fractional anisotropy）value and the ADC(apparent diffusion coefficient) value of relational interesting area（corpus callosum、brainstem、basal ganglia）to analyse the correlation between the FA（fractional anisotropy）value and ADC(apparent diffusion coefficient) value and GCS(Glasgow Coma Scale) and coma time,so that the investigators can quantify the damage degree of patients' white matter fiber.By using fiber tractography the investigators can have the extent of recovery of the patient of DAI（diffuse axonal injury） in real-time detection and give guidance for the clinical decision and the judgement of prognosis).

DETAILED DESCRIPTION:
The investigators will examine 15 patients who was firstly diagnosed as diffuse axonal injury and 15 patients negative for magnetic resonance examination with no trauma with DTI(diffusion tensor imaging). The investigators then determine the FA（fractional anisotropy）value and the ADC(apparent diffusion coefficient) value of relational interesting area（corpus callosum、brainstem、basal ganglia）to analyse the correlation between the FA（fractional anisotropy）value and ADC(apparent diffusion coefficient) value and GCS(Glasgow Coma Scale) and coma time,so that the investigators can quantify the damage degree of patients' white matter fiber.At the same time the investigators rebuild the white matter fiber tract(corpus callosum 、corticospinal tract、optic radiation) of patients using diffusion tensor tractography so that the investigators can judge intuitively the extent of damage and recovery. The investigators Trace the repair of nerve fibers after treatment and guide the further treatment.This trial can exactly determine the relationship between the FA（fractional anisotropy）value and ADC(apparent diffusion coefficient) value in relational interesting area and the extent of damage in patient of DAI（diffuse axonal injury）.Meanwhile the trial confirms that the DTI(diffusion tensor imaging) can exactly judge the prognosis of DAI（diffuse axonal injury）.Obviously by using fiber tractography the investigators can have the extent of recovery of the patient of DAI（diffuse axonal injury） in real-time detection and give guidance for the clinical decision and the judgement of prognosis).

ELIGIBILITY:
Inclusion Criteria:

* Has a history of trauma exactly
* Immediate coma after injury
* Increased intracranial pressure level do not agree with clinical illness severity
* No significant changes of CT while with severe clinical manifestations

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient who attend to be diagnosed as diffuse axonal injury with closed craniocerebral injury caused by a traffic accident or a fall injury)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in FA(fractional anisotropy) | Change from FA(fractional anisotropy) within 2 weeks

SECONDARY OUTCOMES:
Change in ADC(apparent diffusion coefficient) | Change from ADC(apparent diffusion coefficient) within 2 weeks

IPD SHARING:
Plan to Share IPD: Yes